CLINICAL TRIAL: NCT06679595
Title: Transmural Care for Chronically Ill Children: Scientific Guidance and Evaluation of Pilot Projects
Acronym: PETRACA
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Centre Hospitalier Regional de la Citadelle (Unknown); Centre Hospitalier Jolimont-Lobbes (Unknown); University Hospital, Antwerp (Other); Universitaire Ziekenhuizen KU Leuven (Other); Centre Hospitalier Universitaire de Liege (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); Universitair Ziekenhuis Brussel (Other); Institut de Pathologie et de Génétique Charleroi (Other); CHC Montlegia (Other); Hôpital universitaire des enfant Reine Fabiola (Unknown)
Responsible Party: Sponsor
Other Study IDs: B670204000193
Record Dates: First submitted 2024-10-09; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Chronic Diseases in Children; Chronic Diseases in Adolescence; Health Personnel; Parents
Keywords: Realist Evaluation; Chronic Disease; Child; Adolescent; Infant; Home Care Services, Hospital-Based
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Children: Children up to the age of 18 with a chronic condition included in a pilot project for paediatric transmural care
  Interventions: Other: Pilot project paediatric transmural care
- Parents: Parents/ legal guardians of children included in a pilot project for paediatric transmural care
  Interventions: Other: Pilot project paediatric transmural care
- Healthcare professionals: Project coordinators and healtcare professionals involved in a pilot project for paediatric transmural care
  Interventions: Other: Pilot project paediatric transmural care

INTERVENTIONS:
Other: Pilot project paediatric transmural care — The implementation of pilot projects for transmural care for chronically ill children

SUMMARY:
The goal of this Realist Evaluation is to evaluate the implementation of pilot projects for transmural care in chronically ill children.

The main question it aims to answer is: To what extent and how do the pilot projects for transmural care for chronically ill children provide an answer to the quintuple aim?

Participants will

* Complete questionnaires at three timepoints
* Participate in focus group interviews

DETAILED DESCRIPTION:
Introduction Chronic diseases have been increasing over the past few years, including in children. The chronic condition affects their daily functioning and quality of life and leads to frequent hospital admissions. To avoid unneccessary hospital admissions and to offer alternative and innovative forms of care, the Belgian Federal Public Service of Public Health, Food Chain Safety and Environment selected five pilot projects for transmural care for chronically ill children. This study was designed to evaluate these projects.

Methods and design The overall approach is a two-year longitudinal prospective Realist Evaluation using a mixed-methods design.

The quantitative strand, using routine data and questionnaires, will examine whether data from children, parents/legal guardians and healthcare professionals involved in a pilot project for paediatric transmural care comply with the quintuple aim outcomes.

The qualitative strand will be used (1) to evaluate the structure of the interventions, (2) for process evaluation and context analysis, and (3) to gather more in-depth information. This includes document analysis (including logbooks), focus groups with children, parents/legal guardians and healthcare professionals, and non-participatory observations.

Ethical Informed consent is required prior to inclusion in the evaluation study. Informed assent is requested from children older than 12 years. For this study, advice is asked from the Research Ethics Committee of Ghent University Hospital

ELIGIBILITY:
Inclusion Criteria:

* Children: any child up to the age of 18 participating in a pilot project for paediatric transmural care.
* Parent/Legal guardian: any parent or legal guardian of a child participating in a pilot project for paediatric transmural care
* Healthcare professionals: any healthcare professional with patient contact involved within a pilot project for paediatric transmural care
* Coordinators: all study and care coordinators involved within a pilot project for paediatric transmural care

Exclusion Criteria:

* No signed informed consent form available

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The setting of the study is defined as the five pilot projects for paediatric transmural care, conducted by Belgian acute care hospitals in collaboration with primary care. These projects focus on transfusions of concentrated red blood cells at home, ventilation of children with a respiratory disease at home, home enzyme therapy by infusion for children suffering from lysosomal metabolic disease and early discharge of neonates with (partial) tube feeding.
  The study population consists of the people for whom the services offered by the pilot project are intended as defined in the implementation plan. This study population can be divided into four subgroups: the patients (children), their parents/legal guardians, healthcare professionals involved and the coordinators of the pilot projects.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | Baseline, 6 months and through study completion, up to 18 months maximum.
  Quality of Life is used as an indicator for the aim "health status". The PedsQL (Paediatric Quality of Life Inventory) 4.0 Generic Core Scales is used to measure health-related quality of life in children and adolescents ages 2 to 18.
  The scale consists of 23 items and has a child self-report and parallel proxy-report format for ages 5-7, 8-12 and 13-18 years. The items are scored on a five-point Likert-scale, ranging from "never a problem" to "almost always a problem";.
Parental Quality of Life | Baseline, 6 months and through study completion, up to 18 months maximum.
  Quality of Life is used as an indicator for the aim "health status". To estimate parent's quality of life, the take care tool (4 domains, 16 items) is used. The items are scored on a three-point Likert-scale, ranging from "Satisfied" to "Not satisfied".
Caregiver burden | Baseline, 6 months and through study completion, up to 18 months maximum.
  Caregiver burden is used as an indicator for the aim "health status". The 4-item version of the Zarit Burden Interview is used to estimate the caregiver burden for the parents. The items are scored on a five-point Likert-scale, ranging from "Never" tot "Nearly Always"
Diagnosis | Through study completion, up to 18 months maximum.
  The diagnosis and date of diagnosis of the participant are collected as an indicator for the aim "health status".
  These data will be extracted from the (electronic) patient records.
Length of stay in the hospital | Through study completion, up to 18 months maximum.
  The length of stay in the hospital, prior to the start of the transmural care of the participant are collected as an indicator for the aim "health status".
  These data will be extracted from the (electronic) patient records.
Length of stay in transmural care | Through study completion, up to 18 months maximum.
  The length of stay in transmural care, measured by counting the total number of days each child receives this care, is an indicator for the aim "health status".
  These data will be extracted from the (electronic) patient records.
Transmural care at school | Through study completion, up to 18 months maximum.
  If transmural care has been given at school, was evaluated as an indicator for the aim "health status".
  These data will be extracted from the (electronic) patient records.
Adverse events | Continuous data collection, until study completion (18 months)
  Adverse events are logged as an indicator for the aims "health status" and "quality of care".
  Adverse events are continuously logged by the project coordinators in a self-developed questionnaire.
Patient experience | Baseline, 6 months and through study completion, up to 18 months maximum.
  Patient experience is used as an indicator for the aim "quality of care". Patient experience is measured among children (or by proxy under the age of 8) and among their parents. To avoid lengthy statements, a questionnaire was developed by the researchers for this purpose. The items are scored on a five-point Likert-scale, ranging from "Strongly disagree" to "Strongly agree".
Parental Empowerment | Baseline, 6 months and through study completion, up to 18 months maximum.
  Parental empowerment is used as an indicator for the aim "quality of care". Patient empowerment is the patient's ability to have control over their health and their ability to be involved in care. In paediatrics, parents advocate strongly for what they feel is best for their child and family and want to feel they are able to make disicions. Therefore, the empowerment of parents is questioned.
  A questionnaire was developed by the researchers for this purpose. The items are scored on a five-point Likert-scale, ranging from "Strongly disagree" to "Strongly agree".
Job Satisfaction | Baseline, 6 months and through study completion, up to 18 months maximum.
  Job Satisfaction is used as an indicator for the aim "value healthcare professionals".
  The Michigan Organizational Assessment Questionnaire Job Satisfaction Subscale (MOAQ-JSS) is used to measure job satisfaction among the healthcare professionals involved. The three items are scored on a five-point Likert-scale, ranging from "Strongly disagree" to "Strongly agree".
Work-related stress | Baseline, 6 months and through study completion, up to 18 months maximum .
  Work-related stress is used as an indicator for the aim "value healthcare professionals".
  Work-related stress is measured using a single question developed by the researchers. The item is scored on a five-point Likert-scale, ranging from "Strongly disagree" to "Strongly agree".
Quality of Work | Baseline, 6 months and through study completion, up to 18 months maximum.
  Quality of Work is used as an indicator for the aim "value healthcare professionals".
  The dimension Quality of Work of the COPSOQ II is used to measure the experience by the healthcare professional of the immediate output of work. The two items are scored on a five-point Likert-scale, ranging from "To a very large extent" to "To a very small extent".
Competence and Training | Baseline, 6 months and through study completion, up to 18 months maximum.
  Competence and Training is used as an indicator for the aim "value healthcare professionals".
  It is important that the healthcare professional providing care at home with children has solid paediatric competencies and experience. Competence and training are questioned among healthcare professionals, using a self-developed questionnaire.
Socio-demographic variables | Baseline, 6 months and through study completion, up to 18 months maximum.
  Socio-demographic variables are used as an indicator for the aim "equity and inclusion".
  These variables are questioned among parents and healthcare professionals.
Socio-economic variables | Baseline, 6 months and through study completion, up to 18 months maximum.
  Socio-economic variables are used as an indicator for the aim "equity and inclusion".
  Financial status, education, employment status and productivity loss based on the iCPQ are questioned among parents.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Van daele, Prof. dr., Principal Investigator — University Hospital, Ghent; Veerle Duprez, dr., Principal Investigator — University Hospital, Ghent
Locations (11):
- Belgium (11):
  - Hôpital universitaire des enfants Reine Fabiola, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Institut de Pathologie et de Génétique Charleroi, Charleroi
  - University Hospital Antwerp, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Brussel, Jette
  - Centre Hospitalier Jolimont-Lobbes, La Louvière
  - Universitaire Ziekenhuizen Leuven, Leuven
  - Centre Hospitalier Régional de la Citadelle, Liège
  - Centre Hospitaliere Universitaire de Liège, Liège
  - Clinique CHC MontLégia, Liège

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dequeker S, Vanderwee K, Van Daele S, Duprez V; PETRACA Study Group. Realist evaluation of Belgian pilot projects for paediatric transmural care: protocol for a mixed methods study. BMJ Open. 2025 Jun 25;15(6):e102152. doi: 10.1136/bmjopen-2025-102152. PMID 40562551